CLINICAL TRIAL: NCT03089294
Title: Low Intensity Extracorporeal Shock Wave Treatment Patients With Vasculogenic Erectile Dysfunction: Standardisation of Treatment Protocol
Brief Title: Low Intensity Extracorporeal Shock Wave Treatment for Erectile Dysfunction: Standardisation of Treatment Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13771/2016
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Low intensity extracorporeal shock wave treatment
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): Patients will receive 2 sessions of LI-ESWT per week for a 6 week period with energy level 4 (12 sessions totally)
  Interventions: Device: Aries ED device
- Group B (Active Comparator): Patients will receive 3 sessions of LI-ESWT per week for a 4 week period with energy level 4 (12 sessions totally)
  Interventions: Device: Aries ED device
- Group C (Active Comparator): Patients will receive 2 sessions of LI-ESWT per week for a 6 week period with energy level 7 (12 sessions totally)
  Interventions: Device: Aries ED device
- Group D (Active Comparator): Patients will receive 3 sessions of LI-ESWT per week for a 4 week period with energy level 7 (12 sessions totally)
  Interventions: Device: Aries ED device

INTERVENTIONS:
Device: Aries ED device — The Dornier Aries-ED device will be used for the purpose of the study. LI-ESWT will be applied to the penile shaft 3 areas, and the 2 crura (two sites)

SUMMARY:
The present study aims to identify the efficacy saturation effect of low intensity extracorporeal shockwave treatment (LI-ESWT) using Aries ED device in men with mild-moderate and severe vasculogenic ED, who have previously responded to oral PDE5-Is. The efficacy and safety of 4 different session frequency protocols will be compared.

DETAILED DESCRIPTION:
This is a randomized, 4 parallel arms, clinical trial with an 18-month recruitment period. All patients will be PDE5I users/responders. After 1 month wash-out period, ED patients will be screened, in order to randomize 96 men with vasculogenic ED, an International Index of Erectile Function ED (IIEF-ED) domain score between 6-25 and abnormal penile triplex-based hemodynamic parameters (peak flow velocity <35cm/sec) in the last 6 months. Additionally, they will be asked to complete the SEP diaries. Patients will be randomized to receive shockwave treatments (12 sessions for all subjects), either twice a week (total of 6 weeks) or three times a week (total of 4 weeks) at energy level 4 or 7, without treatment interval.

Study visits and duration

Visit 1 (day 0): the basic work-up will take place, including medical and sexual history, as well as necessary lab tests, if needed. One month wash-out period will follow. During this period, all subjects will be asked to avoid any drug related to ED (PDE5i) and have at least 2-4 attempts for intercourse. Furthermore, patients will undergo triplex ultrasonography, unless they have already done so in the last 6 months.Also penile dimensions in both flaccid and erect state will be measured.

Visit 2 (day 28 + 3 days): all patients will complete the IIEF-ED domain and will be randomized to one of the four parallel study groups, using an online program. Groups A and C will receive treatment twice per week, at energy level 4 and 7 respectively. Groups B and D will receive treatment three times per week, at energy level 4 and 7 respectively. PDE5i use is prohibited throughout the study.

Treatment Visits: There will be 12 active treatment visits for all 4 Groups. Patients will receive LI-ESWT, according to the study protocol. Interval between 2 treatments will be 3+1 days for Groups A and C (twice/week) whereas 1+1 day for Groups B and D (three times/week). At visit 6 and 12 a penile ultrasonography will be conducted in order to check for potential adverse events related to the treatment.

Follow-up visits 1 - 3 (4, 12 ,24 and 48 weeks post treatment): Patients will complete the IIEF-ED questionnaire and return the completed SEP diaries for the last 4 weeks prior to every visit. Visit data will also be recorded (protocol compliance, adverse events). At Week 12, triplex will be performed by the standard protocol. For Week 4 there is a + 3 days visit window, whereas for weeks 12, 24 and 48 there is a + 2 weeks visit window.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate
2. Age >18
3. Presence of vasculogenic erectile dysfunction for at least 6 months
4. Positive response to PDE5i
5. IIEF-ED score > 6 and IIEF score < 26 after wash out of PDE5i
6. Abnormal penile triplex-based hemodynamic parameters (peak flow velocity <35cm/sec)
7. Stable heterosexual relationship for more than 3 months
8. Sexually active and agree to suspend all ED therapy for the duration of study

Exclusion Criteria:

1. Any cause of ED other than vascular related
2. Previous radiation therapy to pelvis
3. History of radical prostatectomy
4. Clinically significant chronic haematological disease
5. Cardiovascular conditions that prevent sexual activity
6. Peyronie's Disease or penile curvature
7. History of heart attack, stroke or any life- threatening arrhythmia within the prior 6 month
8. Anti-androgens oral or injectables androgens
9. Untreated Hypogonadism as demonstrated by abnormal testosterone levels
10. Malignancy within the past 5 years
11. Any unstable medical, psychiatric condition or spinal cord injury
12. Anatomical or neurological abnormalities in the treatment area
13. Use of any treatment for ED within 7 days of screening ( oral medications, vacuum devices, constrictive devices, injections or urethral suppositories)
14. Known allergy to ultrasound gel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
The percent of subjects who achieve clinically important difference (MCID) in the EF domain score of the IIEF | baseline and 6 month follow up visit
  MCID is defined according to baseline ED severity as:
  * Improvement by 2 or more in the EF domain score of the IIEF for patients with mild ED ( EF scores 17-25) at baseline.
  * Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED(EF scores 11-16) at baseline
  * Improvement by 7 or more in the EF domain score of the IIEF for patients with severe ED (EF scores 0-10) at baseline

SECONDARY OUTCOMES:
Change in the EF domain score of the IIEF | baseline, 6 month follow up visit and 12 month follow up visit
  EF domain of the IIEF questionnaire will be completed
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline, 6 month follow up visit and 12 month follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
Change in mean peak systolic velocity (PSV) | baseline and 3 month follow up visit
  Mean peak systolic velocity will be measured by penile triplex ultrasonography by the same investigator.
Number of patients with treatment related adverse events | 54 weeks (Group A and Group C), 52 weeks (Group B and Group D)
  Potential treatment related adverse events after the first LI-ESWT session and during the 12 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — Institute for the Study of Urological Diseases (ISUD)
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clavijo RI, Kohn TP, Kohn JR, Ramasamy R. Effects of Low-Intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2017 Jan;14(1):27-35. doi: 10.1016/j.jsxm.2016.11.001. Epub 2016 Dec 13. PMID 27986492
- [Background] Lu Z, Lin G, Reed-Maldonado A, Wang C, Lee YC, Lue TF. Low-intensity Extracorporeal Shock Wave Treatment Improves Erectile Function: A Systematic Review and Meta-analysis. Eur Urol. 2017 Feb;71(2):223-233. doi: 10.1016/j.eururo.2016.05.050. Epub 2016 Jun 16. PMID 27321373
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209
- [Background] Gruenwald I, Kitrey ND, Appel B, Vardi Y. Low-Intensity Extracorporeal Shock Wave Therapy in Vascular Disease and Erectile Dysfunction: Theory and Outcomes. Sex Med Rev. 2013 Jul;1(2):83-90. doi: 10.1002/smrj.9. Epub 2015 Oct 18. PMID 27784587